CLINICAL TRIAL: NCT00862043
Title: Sildenafil for Improving Outcomes After Valvular Correction
Brief Title: Sildenafil for Secondary Pulmonary Hypertension Due to Valvular Disease
Acronym: SIOVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación de Investigación en Red en Enfermedades Cardiovasculares (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIBHGM-SIOVAC; 2007-007033-40 (EudraCT Number); EC07-90772 (Other: Agencia Española del Medicamento y Productos Sanitarios)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Hypertension; Valvular Heart Disease
Keywords: Secondary Pulmonary Hypertension; Valvular Heart Disease; Phosphodiesterase-Inhibitors; Sildenafil; Outcomes Research
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Valve Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil Citrate (Experimental): Sildenafil Citrate 40 mg t.i.d. oral
  Interventions: Drug: Sildenafil Citrate
- Placebo (Placebo Comparator): Sildenafil-matched oral placebo 40 mg t.i.d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — 40 mg t.i.d.
  Arms: Sildenafil Citrate
Drug: Placebo — Placebo t.i.d.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of the mid-term treatment with sildenafil in patients with persistent moderate or severe pulmonary hypertension (PH) after a heart valve intervention.

DETAILED DESCRIPTION:
Phase IV, prospective, multicenter, randomized, double-blind, placebo-controlled, academically funded clinical trial, with 6 months follow-up. A total of 354 patients will be recruited. Inclusion criteria are: 1) successful surgical or percutaneous repair of a cardiac valve at least one year before screening and 2) persistent moderate or severe PH, and 3) absence of any residual significant valvular lesion. Patients will be randomized 1:1 to received sildenafil 40 mg t.i.d. or placebo. The primary endpoint is a clinical composite score combining: all-cause mortality, hospital admission for heart failure, World Health Organization (WHO) functional class, and the patient global assessment score. Additional clinical and mechanistic secondary end-points are defined.

ELIGIBILITY:
Inclusion Criteria:

* Age at the date of selection ≥ 18 years
* Mean pulmonary pressure ≥ 30 mmHg, measured by a Swan-Ganz catheter placed in the pulmonary artery
* Heart valve intervention: surgical or percutaneous replacement, repair or dilatation performed at least one year before inclusion
* Stable clinical condition for at least one month, without hospital admissions for heart failure, and on appropriate and stable doses of conventional cardiovascular medications

Exclusion Criteria:

* Requiring or likely to require the following medications: organic nitrates, alpha-blocker therapy, potent cytochrome P450 3A4 inhibitors (erythromycin, ketoconazole, cimetidine, HIV protease inhibitors such ritonavir and saquinavir) Patients who have suffered a myocardial infarction, stroke, or life-threatening arrhythmia within the last 6 months.
* Patients with resting hypotension, with systolic blood pressure < 90 mmHg
* Patients with retinitis pigmentosa
* Anatomical deformation of the penis (such as angulation, cavernosal fibrosis or Peyronie's disease) or patients who have conditions which may predispose them to priapism (such as sickle cell anemia, multiple myeloma, or leukemia)
* Severe renal impairment with creatinine clearance < 30 ml/min
* Significant hepatic dysfunction
* Prosthesis or valvular dysfunction with hemodynamic repercussion.
* Pregnant or breast-feeding women
* Patients unlikely to cooperate in the study or with inability or unwillingness to give informed consent
* Life expectancy less than 2 years due to non-cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Combined Outcome End-Point: all-cause mortality or hospital admission for heart failure, worsening of World Health Organization (WHO) functional class, or of the patient global assessment score | Six months

SECONDARY OUTCOMES:
Change from baseline to the sixth month in the in the six-minute walk test | 6 Months
Change on WHO functional capacity | 3 & 6 Months
All cause mortality | 6 Months
Cardiovascular mortality | 6 months
Number of hospital admissions caused by or related to heart failure in each patient | 6 months
Rate of progression/regression of tricuspid regurgitation by Doppler-echocardiography | 3 & 6 Months
Change on right ventricular (RV) dimensions and function assessed by Doppler echocardiography | 3 & 6 months
Change on RV volumes and function assessed by cardiac magnetic resonance | 6 Months
Change on the right catheterization hemodynamic parameters | 6 Months
Identify patients who are more likely to respond to therapy by pharmacogenetics analysis | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bermejo, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Maranon
Locations (18):
- Spain (18):
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Alava, Vitoria-Gasteiz, Alava
  - Hospital German Trias y Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu y San Pau, Barcelona, Barcelon
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Juan Canalejo, A Coruña, La Coruna
  - Hospital de Leon, León, Leon
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Infanta Leonor, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital Clínico de Valladolid, Valladolid, Valladolid
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital Virgen de las Nieves, Granada

REFERENCES:
- [Derived] Bermejo J, Gonzalez-Mansilla A, Mombiela T, Fernandez AI, Martinez-Legazpi P, Yotti R, Garcia-Orta R, Sanchez-Fernandez PL, Castano M, Segovia-Cubero J, Escribano-Subias P, Alberto San Roman J, Borras X, Alonso-Gomez A, Botas J, Crespo-Leiro MG, Velasco S, Bayes-Genis A, Lopez A, Munoz-Aguilera R, Jimenez-Navarro M, Gonzalez-Juanatey JR, Evangelista A, Elizaga J, Martin-Moreiras J, Gonzalez-Santos JM, Moreno-Escobar E, Fernandez-Aviles F; SIOVAC ("Sildenafil for Improving Outcomes after VAlvular Correction") Investigators. Persistent Pulmonary Hypertension in Corrected Valvular Heart Disease: Hemodynamic Insights and Long-Term Survival. J Am Heart Assoc. 2021 Jan 19;10(2):e019949. doi: 10.1161/JAHA.120.019949. Epub 2021 Jan 5. PMID 33399006
- [Derived] Bermejo J, Yotti R, Garcia-Orta R, Sanchez-Fernandez PL, Castano M, Segovia-Cubero J, Escribano-Subias P, San Roman JA, Borras X, Alonso-Gomez A, Botas J, Crespo-Leiro MG, Velasco S, Bayes-Genis A, Lopez A, Munoz-Aguilera R, de Teresa E, Gonzalez-Juanatey JR, Evangelista A, Mombiela T, Gonzalez-Mansilla A, Elizaga J, Martin-Moreiras J, Gonzalez-Santos JM, Moreno-Escobar E, Fernandez-Aviles F; Sildenafil for Improving Outcomes after VAlvular Correction (SIOVAC) investigators. Sildenafil for improving outcomes in patients with corrected valvular heart disease and persistent pulmonary hypertension: a multicenter, double-blind, randomized clinical trial. Eur Heart J. 2018 Apr 14;39(15):1255-1264. doi: 10.1093/eurheartj/ehx700. PMID 29281101
- See also: Funding Agent — http://www.mineco.gob.es
- See also: Cardiovascular Research Spanish National Network — http://www.redcardiovascular.com